CLINICAL TRIAL: NCT04016142
Title: Phase II Trial of Weekly Carboplatin-Paclitaxel Adjuvant Chemotherapy After Intensity Modulated Extended-field Chemoradiation in the Treatment of Locally Advanced Cervical Cancer with Para-aortic Positive Nodes
Brief Title: Carboplatin-Paclitaxel Adjuvant Chemotherapy in the Treatment of Locally Advanced Cervical Cancer
Acronym: ACCRAPAN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study is discontinued because of recruitment failure, and for strategic reason (competitive trials with immunotherapy)
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACCRAPAN-1806; 2018-001752-35 (EudraCT Number)
Record Dates: First submitted 2019-05-31; First posted 2019-07-11 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Locally Advanced Cancer; Cervical Cancer
Keywords: Adjuvant Chemotherapy; Cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Chemotherapy, Adjuvant; CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Carboplatin-Paclitaxel adjuvant chemotherapy (Experimental): Patients
  * will be registered in the first part of the study at diagnosis and will receive a first part of treatment corresponding to a standard of care (standard concomitant radio-chemotherapy, "Part 1 of the study").
  * will be included in the second part of the study for the second part of treatment (experimental adjuvant chemotherapy, "Part 2 of the study"), providing they fulfill eligibility criteria at this stage (no progression during Part 1 of the study and no medical contra-indication to the study treatment).
  Interventions: Drug: Carboplatin-Paclitaxel adjuvant chemotherapy

INTERVENTIONS:
Drug: Carboplatin-Paclitaxel adjuvant chemotherapy — Patients will receive a first part of treatment corresponding to a standard of care (standard concomitant radio-chemotherapy, "Part 1 of the study").
  Then, they will be included in the second part of the study for the second part of treatment (experimental adjuvant chemotherapy, "Part 2 of the study"), providing they fulfill eligibility criteria at this stage.
  The second part consists in 4 cycles of Carboplatin-Paclitaxel adjuvant chemotherapy (one cycle = 3 weeks of treatment and 1 free-week)
  Other Names: Adjuvant Chemotherapy; Carboplatin-Paclitaxel

SUMMARY:
This is a mutlicentric, open-label non-randomized, national, 2-stage phase II trial to assess efficacy and safety of a weekly Carboplatin-Paclitaxel adjuvant chemotherapy after intensity modulated extended-field chemoradiation in patient suffering from of locally advanced cervical cancer with para-aortic positive nodes.

DETAILED DESCRIPTION:
This is a mutlicentric, open-label non-randomized, national, 2-stage phase II trial to assess efficacy and safety of a weekly Carboplatin-Paclitaxel adjuvant chemotherapy after intensity modulated extended-field chemoradiation in patient suffering from of locally advanced cervical cancer with para-aortic positive nodes.

Patients

* will be registered in the first part of the study at diagnosis and will receive a first part of treatment corresponding to a standard of care (standard concomitant radio-chemotherapy, "Part 1 of the study").
* will be included in the second part of the study for the second part of treatment (experimental adjuvant chemotherapy, "Part 2 of the study"), providing they fulfill eligibility criteria at this stage (no progression during Part 1 of the study and no medical contra-indication to the study treatment).

The primary objective is to evaluate the efficacy of adjuvant chemotherapy with Carboplatin-Paclitaxel administrated in adjuvant situation after concomitant radio-chemotherapy in terms of Progression Free Survival (PFS) in patients treated for a locally advanced cervical cancer presenting positive lombo-aortic lymph nodes.

ELIGIBILITY:
PART 1:

Inclusion Criteria:

* Female patient aged more than 18 years old
* Histological diagnosis of squamous cell carcinoma, adenocarcinoma or adenosquamous cell carcinoma of the cervix
* With locally advanced cervical cancer (FIGO stage IIIC2)
* With para-aortic or iliac common nodes positive on PET-scan or after laparoscopic surgical staging if PET-scan negative
* ECOG Performance Status ≤ 2
* Adequate hematologic function: Absolute Neutrophil Count (ANC) ≥ 1,500/mm3, platelets ≥ 100,000/mm3, hemoglobin ≥ 10g/dL
* Adequate renal function: creatinine clearance (estimated according to MDRD formula) ≥ 60ml/min/1.73m²
* Adequate hepatic function: Aspartate aminotransferase (ALT)/ Alanine aminotransferase (ALT) ≤ 2.5 × upper normal limit (UNL); Total bilirubin ≤ 1.5 x UNL (except in case of Gilbert's disease)
* Negative serum pregnancy test within 7 days prior to treatment for women of childbearing potential. For non-menopaused women, if not surgically sterilized, willing to accept the use of an effective contraceptive regimen during the treatment period and at least 6 months after the end of treatment
* Absence of contraindication to receive the products used in this study (products used in concomitant/ adjuvant chemotherapy) according to the most recent SmPC of these products (available at http://base-donnees-publique.medicaments.gouv.fr/)
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow-up
* Patient covered by the French "Social Security" regime
* Signed informed consent form

Exclusion Criteria:

* Histological diagnosis of sarcoma
* Previous hysterectomy or planned hysterectomy as part of their initial cervix cancer therapy,
* Presence of distant metastases other than lombo-aortic lymph nodes
* Patient with other invasive malignancies, with the exception of non-melanoma skin cancer, who had (or have) any evidence of the other cancer present within the last 5 years
* Patient with bilateral hydronephrosis unless at least one side has been stented
* Prior diagnosis of Crohn's disease or ulcerative colitis or sclerodermia
* Other uncontrolled intercurrent disease including, but not limited to: active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia
* Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation
* Pregnant or breastfeeding woman,
* Participation in another therapeutic trial with an experimental molecule for the current disease
* Psychiatric illness or social situation that would limit compliance with study requirement, substantially increase the risk of side effects, or compromise the ability of the patient to give written informed consent
* Inability to comply with medical follow-up of the trial (geographical, social or psychic reasons)
* Person under guardianship or curatorship

PART 2:

Inclusion Criteria:

* Maintained consent
* Adequate hematologic function: Absolute Neutrophil Count (ANC) ≥ 1,500/mm3, platelets ≥ 100,000/mm3, hemoglobin ≥ 10g/dL
* Adequate renal function: creatinine clearance (estimated according to MDRD formula) ≥ 60ml/min/1.73m2
* Adequate hepatic function: Aspartate aminotransferase (ALT)/ Alanine aminotransferase (ALT) ≤ 2.5 × upper normal limit (UNL); Total bilirubin ≤ 1.5 x UNL (except in case of Gilbert's disease)
* Patient having received curative intent chemo-radiation therapy with the following recommendations:

  * extended field CT-RT delivered by IMRT: 45-50Gy according the dosimetry limitation histogram dose volume (HDV) in whole pelvis and Para Aortic volumes + concomitant boost on macroscopic nodes defined as PET-positive
  * associated with weekly Cisplatin (40mg/m²)
  * followed by image guided brachytherapy. Patient will be eligible even in case of temporary stop of radiation therapy, provided she has received a total dose of 45Gy and a concomitant boost. Patient should have received at least 3 injections of Cisplatin 40mg/m² during radiation therapy.

Exclusion Criteria:

* Progression during Part 1,
* Contraindication for one of the study drug in particular the residual toxicity of Part 1 (radio-chemotherapy) such as:

  * Renal failure (defined as creatinine clearance according to MDRD formula < 60 mL/ min/1.73m2),
  * Any clinical residual toxicity (including peripheral neuropathy) ≥ grade 2 (as per CTCAE v5),
* Radiation therapy prematurely stopped (total dose on whole pelvis and on nodes not received)
* Cumulative dose of Cisplatin received less than 120 mg/m².

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient has to suffer from a cervical cancer.
Enrollment: 21 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival with adjuvant chemotherapy | From the date of inclusion in the Part 2 of the study until the date of first progression or relapse (local, lymph nodes or metastatic) or death whatever the cause. Assessed up to 64 months.
  To evaluate the efficacy of adjuvant chemotherapy with Carboplatin-Paclitaxel administrated in adjuvant situation after concomitant radio-chemotherapy in terms of Progression Free Survival (PFS) in patients treated for a locally advanced cervical cancer presenting positive lombo-aortic lymph nodes.
  Progression will be based on a MRI scan, done during the usual oncologic follow-up: every 3 months during the 2 first years after radio-chemotherapy, and then every 6 months during 3 years.
  Progression will be evaluated with RECIST criteria v1.1. The main analysis of this phase II trial will focus on the 2-year PFS rate from inclusion in the Part 2, but the whole curve will be estimated.

SECONDARY OUTCOMES:
Overall Survival with adjuvant chemotherapy | From the date of inclusion in the Part 2 of the study until the date of death whatever the cause. Assessed up to 64 months.
  To evaluate efficacy of adjuvant chemotherapy with Carboplatin-Paclitaxel in terms of Overall Survival (OS) in patients treated for a locally advanced cervical cancer presenting positive lombo-aortic lymph nodes.
  OS will be estimated with the Kaplan-Meier method.
Metastasis Free Survival with adjuvant chemotherapy | From the date of inclusion in the Part 2 of the study until the date of first metastatic progression or death whatever the cause. Assessed up to 64 months.
  To evaluate efficacy of adjuvant chemotherapy with Carboplatin-Paclitaxel in terms of Metastasis Free Survival (MFS) in patients treated for a locally advanced cervical cancer presenting positive lombo-aortic lymph nodes.
  Metastatic progressions will be evaluated with the RECIST criteria.
Number of Cycles Received of adjuvant chemotherapy | From the date of inclusion in the Part 2 of the study until the date of adjuvant chemotherapy ending or patient study output or death whatever the cause. Up to 4 months.
  To describe feasibility of adjuvant chemotherapy in terms of number of cycles received, separately for each molecule Carboplatin and Paclitaxel.
  The number of cycles will be recorded in the data base with the date and doses of injections, allowing the calculation of the Relative Dose Intensity.
  Reasons of treatment stop or dose modification will also be recorded.
Progression Free Survival with concomitant chemo-radiotherapy associated to brachytherapy | From the date of inclusion in the Part 1 of the study until the date of first progression or relapse (local, lymph nodes or metastatic) or death whatever the cause. Assessed up to 67 months.
  To evaluate the efficacy of adjuvant chemotherapy with concomitant chemo-radiotherapy associated to brachytherapy in terms of Progression Free Survival (PFS) in patients treated for a locally advanced cervical cancer presenting positive lombo-aortic lymph nodes.
  Progression will be based on a MRI scan, done during the usual oncologic follow-up: every 3 months during the 2 first years after radio-chemotherapy, and then every 6 months during 3 years.
  Progression will be evaluated with RECIST criteria v1.1.
Overall Survival with concomitant chemo-radiotherapy associated to brachytherapy | From the date of inclusion in the Part 1 of the study until the date of death whatever the cause. Assessed up to 67 months.
  To evaluate efficacy of concomitant chemo-radiotherapy associated to brachytherapy in terms of Overall Survival (OS) in patients treated for a locally advanced cervical cancer presenting positive lombo-aortic lymph nodes.
  OS will be estimated with the Kaplan-Meier method.
Metastasis Free Survival with concomitant chemo-radiotherapy associated to brachytherapy | From the date of inclusion in the Part 1 of the study until the date of first metastatic progression or death whatever the cause. Assessed up to 67 months.
  To evaluate efficacy of concomitant chemo-radiotherapy associated to brachytherapy in terms of Metastasis Free Survival (MFS) in patients treated for a locally advanced cervical cancer presenting positive lombo-aortic lymph nodes.
  Metastatic progressions will be evaluated with the RECIST criteria.
Number of Cycles Received of concomitant chemo-radiotherapy associated to brachytherapy | From the date of inclusion in the Part 1 of the study until the date of concomitant chemo-radiotherapy associated to brachytherapy ending or patient study output or death whatever the cause. Assessed up to 12 weeks.
  To describe feasibility of the concomitant chemo-radiotherapy associated to brachytherapy (Part 1 of the study) in terms of number of cycles received.
  The number of cycles will be recorded in the data base with the date and doses of injections, allowing the calculation of the Relative Dose Intensity.
  Reasons of treatment stop or dose modification will also be recorded.
Safety of the whole treatment | From the date of inclusion in the Part 1 of the study, up to 5 years after the end of radiation therapy or until progression (whichever occurs first).
  To describe safety of the whole treatment (part 1 & 2) in terms of Adverse Event.
  During the first part of the study (concomitant radio-chemotherapy), all AE (Adverse Events) will be reported. AE occurring after end of treatment will not be collected for patients withdrawn from the study at the end of the first part. For the second part of the study (adjuvant chemotherapy), all AE will be reported up to 30 days after the end of adjuvant chemotherapy, until progression if any. Then, only AE possibly related to chemotherapy or radiation therapy will be collected, up to 5 years after the end of radiation therapy or until progression (whichever occurs first). All AE will be graded using the NCI-CTCAE v5.0 and AE of grade >2 will be considered as severe AE.

CONTACTS AND LOCATIONS:
Overall Officials: Florence Le Tinier, MD, Principal Investigator — Centre Oscar Lambret
Locations (6):
- France (6):
  - Centre Marie Curie, Arras, France
  - Centre Pierre Curie, Beuvry, France
  - Centre Léonard de Vinci, Dechy, France
  - Centre Oscar Lambret, Lille, France
  - Clinique des dentellières, Valenciennes, France
  - Centre Hospitalier de Lens, Lens

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shayne M, Crawford J, Dale DC, Culakova E, Lyman GH; ANC Study Group. Predictors of reduced dose intensity in patients with early-stage breast cancer receiving adjuvant chemotherapy. Breast Cancer Res Treat. 2006 Dec;100(3):255-62. doi: 10.1007/s10549-006-9254-4. Epub 2006 May 17. PMID 16705366
- [Background] Chemoradiotherapy for Cervical Cancer Meta-Analysis Collaboration. Reducing uncertainties about the effects of chemoradiotherapy for cervical cancer: a systematic review and meta-analysis of individual patient data from 18 randomized trials. J Clin Oncol. 2008 Dec 10;26(35):5802-12. doi: 10.1200/JCO.2008.16.4368. Epub 2008 Nov 10. PMID 19001332
- [Background] Gouy S, Morice P, Narducci F, Uzan C, Gilmore J, Kolesnikov-Gauthier H, Querleu D, Haie-Meder C, Leblanc E. Nodal-staging surgery for locally advanced cervical cancer in the era of PET. Lancet Oncol. 2012 May;13(5):e212-20. doi: 10.1016/S1470-2045(12)70011-6. PMID 22554549
- [Background] Leblanc E, Narducci F, Frumovitz M, Lesoin A, Castelain B, Baranzelli MC, Taieb S, Fournier C, Querleu D. Therapeutic value of pretherapeutic extraperitoneal laparoscopic staging of locally advanced cervical carcinoma. Gynecol Oncol. 2007 May;105(2):304-11. doi: 10.1016/j.ygyno.2006.12.012. Epub 2007 Jan 29. PMID 17258799
- [Background] Grigsby PW. The prognostic value of PET and PET/CT in cervical cancer. Cancer Imaging. 2008 Jul 24;8(1):146-55. doi: 10.1102/1470-7330.2008.0022. PMID 18694852
- [Background] Tsai CS, Chang TC, Lai CH, Tsai CC, Ng KK, Hsueh S, Yen TC, Hong JH. Preliminary report of using FDG-PET to detect extrapelvic lesions in cervical cancer patients with enlarged pelvic lymph nodes on MRI/CT. Int J Radiat Oncol Biol Phys. 2004 Apr 1;58(5):1506-12. doi: 10.1016/j.ijrobp.2003.09.013. PMID 15050330
- [Background] Ahmed RS, Kim RY, Duan J, Meleth S, De Los Santos JF, Fiveash JB. IMRT dose escalation for positive para-aortic lymph nodes in patients with locally advanced cervical cancer while reducing dose to bone marrow and other organs at risk. Int J Radiat Oncol Biol Phys. 2004 Oct 1;60(2):505-12. doi: 10.1016/j.ijrobp.2004.03.035. PMID 15380585
- [Background] Rotman M, Pajak TF, Choi K, Clery M, Marcial V, Grigsby PW, Cooper J, John M. Prophylactic extended-field irradiation of para-aortic lymph nodes in stages IIB and bulky IB and IIA cervical carcinomas. Ten-year treatment results of RTOG 79-20. JAMA. 1995 Aug 2;274(5):387-93. PMID 7616634
- [Background] Eifel PJ, Winter K, Morris M, Levenback C, Grigsby PW, Cooper J, Rotman M, Gershenson D, Mutch DG. Pelvic irradiation with concurrent chemotherapy versus pelvic and para-aortic irradiation for high-risk cervical cancer: an update of radiation therapy oncology group trial (RTOG) 90-01. J Clin Oncol. 2004 Mar 1;22(5):872-80. doi: 10.1200/JCO.2004.07.197. PMID 14990643
- [Background] Morris M, Eifel PJ, Lu J, Grigsby PW, Levenback C, Stevens RE, Rotman M, Gershenson DM, Mutch DG. Pelvic radiation with concurrent chemotherapy compared with pelvic and para-aortic radiation for high-risk cervical cancer. N Engl J Med. 1999 Apr 15;340(15):1137-43. doi: 10.1056/NEJM199904153401501. PMID 10202164
- [Background] Grigsby PW, Heydon K, Mutch DG, Kim RY, Eifel P. Long-term follow-up of RTOG 92-10: cervical cancer with positive para-aortic lymph nodes. Int J Radiat Oncol Biol Phys. 2001 Nov 15;51(4):982-7. doi: 10.1016/s0360-3016(01)01723-0. PMID 11704321
- [Background] Mundt AJ, Mell LK, Roeske JC. Preliminary analysis of chronic gastrointestinal toxicity in gynecology patients treated with intensity-modulated whole pelvic radiation therapy. Int J Radiat Oncol Biol Phys. 2003 Aug 1;56(5):1354-60. doi: 10.1016/s0360-3016(03)00325-0. PMID 12873680
- [Background] Cihoric N, Tapia C, Kruger K, Aebersold DM, Klaeser B, Lossl K. IMRT with (1)(8)FDG-PET\CT based simultaneous integrated boost for treatment of nodal positive cervical cancer. Radiat Oncol. 2014 Mar 25;9:83. doi: 10.1186/1748-717X-9-83. PMID 24661323
- [Background] Vargo JA, Kim H, Choi S, Sukumvanich P, Olawaiye AB, Kelley JL, Edwards RP, Comerci JT, Beriwal S. Extended field intensity modulated radiation therapy with concomitant boost for lymph node-positive cervical cancer: analysis of regional control and recurrence patterns in the positron emission tomography/computed tomography era. Int J Radiat Oncol Biol Phys. 2014 Dec 1;90(5):1091-8. doi: 10.1016/j.ijrobp.2014.08.013. Epub 2014 Oct 8. PMID 25303889
- [Background] Perry LJ, Mathews C, Nugent E, Farrell R, Zorn K, Moore K. Outcomes of cervical cancer and positive para-aortic lymph nodes in the modern era of chemoradiation. Int J Gynecol Cancer. 2014 Mar;24(3):564-9. doi: 10.1097/IGC.0000000000000093. PMID 24552890
- [Background] Gouy S, Morice P, Narducci F, Uzan C, Martinez A, Rey A, Bentivegna E, Pautier P, Deandreis D, Querleu D, Haie-Meder C, Leblanc E. Prospective multicenter study evaluating the survival of patients with locally advanced cervical cancer undergoing laparoscopic para-aortic lymphadenectomy before chemoradiotherapy in the era of positron emission tomography imaging. J Clin Oncol. 2013 Aug 20;31(24):3026-33. doi: 10.1200/JCO.2012.47.3520. Epub 2013 Jul 15. PMID 23857967
- [Background] Duenas-Gonzalez A, Zarba JJ, Patel F, Alcedo JC, Beslija S, Casanova L, Pattaranutaporn P, Hameed S, Blair JM, Barraclough H, Orlando M. Phase III, open-label, randomized study comparing concurrent gemcitabine plus cisplatin and radiation followed by adjuvant gemcitabine and cisplatin versus concurrent cisplatin and radiation in patients with stage IIB to IVA carcinoma of the cervix. J Clin Oncol. 2011 May 1;29(13):1678-85. doi: 10.1200/JCO.2009.25.9663. Epub 2011 Mar 28. PMID 21444871
- [Background] Mabuchi S, Morishige K, Fujita M, Tsutsui T, Sakata M, Enomoto T, Kimura T. The activity of carboplatin and paclitaxel for recurrent cervical cancer after definitive radiotherapy. Gynecol Oncol. 2009 May;113(2):200-4. doi: 10.1016/j.ygyno.2009.02.008. Epub 2009 Mar 6. PMID 19268342
- [Background] Tinker AV, Bhagat K, Swenerton KD, Hoskins PJ. Carboplatin and paclitaxel for advanced and recurrent cervical carcinoma: the British Columbia Cancer Agency experience. Gynecol Oncol. 2005 Jul;98(1):54-8. doi: 10.1016/j.ygyno.2005.03.037. PMID 15904950
- [Background] Mabuchi S, Morishige K, Enomoto T, Kimura T. Carboplatin and paclitaxel as an initial treatment in patients with stage IVb cervical cancer: a report of 7 cases and a review of the literature. J Gynecol Oncol. 2010 Jun;21(2):93-6. doi: 10.3802/jgo.2010.21.2.93. Epub 2010 Jun 30. PMID 20613898
- [Background] Neoadjuvant Chemotherapy for Locally Advanced Cervical Cancer Meta-analysis Collaboration. Neoadjuvant chemotherapy for locally advanced cervical cancer: a systematic review and meta-analysis of individual patient data from 21 randomised trials. Eur J Cancer. 2003 Nov;39(17):2470-86. doi: 10.1016/s0959-8049(03)00425-8. PMID 14602133
- [Background] McCormack M, Kadalayil L, Hackshaw A, Hall-Craggs MA, Symonds RP, Warwick V, Simonds H, Fernando I, Hammond M, James L, Feeney A, Ledermann JA. A phase II study of weekly neoadjuvant chemotherapy followed by radical chemoradiation for locally advanced cervical cancer. Br J Cancer. 2013 Jun 25;108(12):2464-9. doi: 10.1038/bjc.2013.230. Epub 2013 May 21. PMID 23695016
- [Background] Sparano JA, Wang M, Martino S, Jones V, Perez EA, Saphner T, Wolff AC, Sledge GW Jr, Wood WC, Davidson NE. Weekly paclitaxel in the adjuvant treatment of breast cancer. N Engl J Med. 2008 Apr 17;358(16):1663-71. doi: 10.1056/NEJMoa0707056. PMID 18420499
- [Background] ELLIS RE. The distribution of active bone marrow in the adult. Phys Med Biol. 1961 Jan;5:255-8. doi: 10.1088/0031-9155/5/3/302. No abstract available. PMID 13726497
- [Background] Vande Berg BC, Malghem J, Lecouvet FE, Maldague B. Magnetic resonance imaging of the normal bone marrow. Skeletal Radiol. 1998 Sep;27(9):471-83. doi: 10.1007/s002560050423. PMID 9809875
- [Background] Platta CS, Bayliss A, McHaffie D, Tome WA, Straub MR, Bradley KA. A dosimetric analysis of tomotherapy based intensity modulated radiation therapy with and without bone marrow sparing in gynecologic malignancies. Technol Cancer Res Treat. 2013 Feb;12(1):19-29. doi: 10.7785/tcrt.2012.500300. Epub 2012 Sep 10. PMID 22974331
- [Background] Mell LK, Kochanski JD, Roeske JC, Haslam JJ, Mehta N, Yamada SD, Hurteau JA, Collins YC, Lengyel E, Mundt AJ. Dosimetric predictors of acute hematologic toxicity in cervical cancer patients treated with concurrent cisplatin and intensity-modulated pelvic radiotherapy. Int J Radiat Oncol Biol Phys. 2006 Dec 1;66(5):1356-65. doi: 10.1016/j.ijrobp.2006.03.018. Epub 2006 Jun 6. PMID 16757127
- [Background] Chang Y, Yang ZY, Li GL, Li Q, Yang Q, Fan JQ, Zhao YC, Song YQ, Wu G. Correlations Between Radiation Dose in Bone Marrow and Hematological Toxicity in Patients With Cervical Cancer: A Comparison of 3DCRT, IMRT, and RapidARC. Int J Gynecol Cancer. 2016 May;26(4):770-6. doi: 10.1097/IGC.0000000000000660. PMID 26844613
- [Background] Yang TJ, Oh JH, Apte A, Son CH, Deasy JO, Goodman KA. Clinical and dosimetric predictors of acute hematologic toxicity in rectal cancer patients undergoing chemoradiotherapy. Radiother Oncol. 2014 Oct;113(1):29-34. doi: 10.1016/j.radonc.2014.09.002. Epub 2014 Oct 7. PMID 25304718
- [Background] Lujan AE, Mundt AJ, Yamada SD, Rotmensch J, Roeske JC. Intensity-modulated radiotherapy as a means of reducing dose to bone marrow in gynecologic patients receiving whole pelvic radiotherapy. Int J Radiat Oncol Biol Phys. 2003 Oct 1;57(2):516-21. doi: 10.1016/s0360-3016(03)00521-2. PMID 12957265
- [Background] Lim K, Small W Jr, Portelance L, Creutzberg C, Jurgenliemk-Schulz IM, Mundt A, Mell LK, Mayr N, Viswanathan A, Jhingran A, Erickson B, De los Santos J, Gaffney D, Yashar C, Beriwal S, Wolfson A, Taylor A, Bosch W, El Naqa I, Fyles A; Gyn IMRT Consortium. Consensus guidelines for delineation of clinical target volume for intensity-modulated pelvic radiotherapy for the definitive treatment of cervix cancer. Int J Radiat Oncol Biol Phys. 2011 Feb 1;79(2):348-55. doi: 10.1016/j.ijrobp.2009.10.075. Epub 2010 May 14. PMID 20472347
- [Background] A'Hern RP. Sample size tables for exact single-stage phase II designs. Stat Med. 2001 Mar 30;20(6):859-66. doi: 10.1002/sim.721. PMID 11252008